CLINICAL TRIAL: NCT02072590
Title: Improved Diagnostics of Celiac Disease in Children
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Other Study IDs: R11187
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Celiac Disease; Eosinophilic Esophagitis
Keywords: Celiac disease; Eosinophilic esophagitis; Endomysial antibodies; Transglutaminase antibodies; Small-bowel
MeSH Terms: conditions — Celiac Disease; Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, intestinal mucosal biopsies
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purpose of this study is to improve the diagnostics of celiac disease and reduce the need for invasive endoscopic studies in children. Further, the investigators aim to investigate the natural history and risk of complications in children with celiac disease or gluten sensitivity and to create a large scientific database.

DETAILED DESCRIPTION:
Prevalence of celiac disease is on a steep rise in Western countries, but due to difficult diagnosis the majority of patients remain unrecognized. Undiagnosed celiac disease causes incremental burden to the health care and predisposes to severe complications. On the other hand, increasing screening in at-risk groups of celiac disease frequently detects seropositive subjects with no obvious symptoms and/or still normal small-bowel mucosal morphology. At present the natural history and benefits of an early diagnosis in such individuals is poorly known. Further, the endoscopic demonstration of the small-intestinal damage required for the diagnosis is unpleasant, expensive and often misleading. New serology-based diagnostic criteria have been suggested but prospective data is lacking. Aims of the present study are to improve the diagnostic yield and accuracy of the current diagnostic methods and to develop novel non-invasive methods and biomarkers for early detection of celiac disease. In addition, the investigators will evaluate natural history of celiac disease in screening-detected asymptomatic children and in those with positive serology but normal histology, and form a large database for future clinical and translational studies. The study and patient collection are to be conducted at the pediatric clinics in Finland and in Romania. All children referred due to suspicion of celiac disease or gluten sensitivity will be asked to participate to the study. Patient samples and clinical information are collected during the routine visits and the study does not include any additional visits or endoscopies. The total duration of the study is 10 years but data will be analyzed on-line.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of celiac disease or gluten sensitivity
* Age below 18 years

Exclusion Criteria:

* Study refusal
* Age 18 years or more

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospital clinic; secondary and tertiary centers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-08; Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Transglutaminase 2 antibodies | Baseline and after 3 months, 6 months and 1 year on a gluten-free diet
  Change of the transglutaminase 2 antibody levels on a gluten-free diet

SECONDARY OUTCOMES:
Serum endomysial antibodies | Baseline and after 3 months, 6 months and 1 year on a gluten-free diet
  Change of the endomysial antibody levels on a gluten-free diet
Visual Analog Scale | Baseline and after 3 months, 6 months and 1 year on a gluten-free diet
  Change in the the subjective perception of health measured by Visual Analog Scale
Dietary compliance | After 3 months, 6 months and 1 year on a gluten-free diet
  Adherence to the gluten-free diet
Height | Baseline and after 3 months, 6 months and 1 year on a gluten-free diet
  Change of height (centimeters) on a gluten-free diet
Weight | Baseline and after 3 months, 6 months and 1 year on a gluten-free diet
  Change of weight (kilograms) on a gluten-free diet

CONTACTS AND LOCATIONS:
Overall Officials: Kalle Kurppa, MD, Principal Investigator — Tampere Centre for Child Health Research, University of Tampere and Tampere University hospital
Locations (2):
- Tampere Centre for Child Health Research, University of Tampere and Tampere University hospital, Tampere, Finland
- University of Medicine and Pharmacy "Carol Davila", Bucharest, Romania, Bucharest, Romania

REFERENCES:
- [Background] Kurppa K, Ashorn M, Iltanen S, Koskinen LL, Saavalainen P, Koskinen O, Maki M, Kaukinen K. Celiac disease without villous atrophy in children: a prospective study. J Pediatr. 2010 Sep;157(3):373-80, 380.e1. doi: 10.1016/j.jpeds.2010.02.070. Epub 2010 Apr 18. PMID 20400102
- [Background] Popp A, Mihu M, Munteanu M, Ene A, Dutescu M, Colcer F, Raducanu D, Laurila K, Anca I, Maki M. Prospective antibody case finding of coeliac disease in type-1 diabetes children: need of biopsy revisited. Acta Paediatr. 2013 Mar;102(3):e102-6. doi: 10.1111/apa.12117. Epub 2013 Jan 4. PMID 23211000
- [Background] Taavela J, Koskinen O, Huhtala H, Lahdeaho ML, Popp A, Laurila K, Collin P, Kaukinen K, Kurppa K, Maki M. Validation of morphometric analyses of small-intestinal biopsy readouts in celiac disease. PLoS One. 2013 Oct 11;8(10):e76163. doi: 10.1371/journal.pone.0076163. eCollection 2013. PMID 24146832
- [Derived] Popp A, Taavela J, Arvola T, Kaukinen K, Maki M, Kurppa K. Bulb biopsies for diagnosing celiac disease in children: A prospective multicenter study using quantitative histomorphometry. J Pediatr Gastroenterol Nutr. 2026 Jan;82(1):129-136. doi: 10.1002/jpn3.70255. Epub 2025 Nov 6. PMID 41195622
- [Derived] Repo M, Lindfors K, Maki M, Huhtala H, Laurila K, Lahdeaho ML, Saavalainen P, Kaukinen K, Kurppa K. Anemia and Iron Deficiency in Children With Potential Celiac Disease. J Pediatr Gastroenterol Nutr. 2017 Jan;64(1):56-62. doi: 10.1097/MPG.0000000000001234. PMID 27101536
- [Derived] Rajalahti T, Repo M, Kivela L, Huhtala H, Maki M, Kaukinen K, Lindfors K, Kurppa K. Anemia in Pediatric Celiac Disease: Association With Clinical and Histological Features and Response to Gluten-free Diet. J Pediatr Gastroenterol Nutr. 2017 Jan;64(1):e1-e6. doi: 10.1097/MPG.0000000000001221. PMID 27035377